CLINICAL TRIAL: NCT02215746
Title: Relative Oral Bioavailability of BI 44370 TA Drinking Solution (100 mg and 200 mg) and BI 44370 TA Tablets (100 mg as Two 50 mg Tablets) With and Without a High Fat Meal in Healthy Male and Female Volunteers: A Single Dose, Open-label, Randomised Six-way Cross-over Trial
Brief Title: Bioavailability of BI 44370 TA Drinking Solution or Tablets With and Without a High Fat Meal in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1246.2
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Solutions

ARMS (6):
- Treatment A (Experimental): BI 44370 TA drinking solution 100 mg fasted
  Interventions: Drug: BI 44370 powder for oral solution
- Treatment B (Experimental): BI 44370 TA drinking solution 100 mg fed
  Interventions: Drug: BI 44370 powder for oral solution; Other: high fat breakfast
- Treatment C (Experimental): BI 44370 TA drinking solution 200 mg fasted
  Interventions: Drug: BI 44370 powder for oral solution
- Treatment D (Experimental): BI 44370 TA drinking solution 200 mg fed
  Interventions: Drug: BI 44370 powder for oral solution; Other: high fat breakfast
- Treatment E (Experimental): 100 mg BI 44370 BS as two tablets 50 mg fasted
  Interventions: Drug: BI 44370 tablet
- Treatment F (Experimental): 100 mg BI 44370 BS as two tablets 50 mg fed
  Interventions: Drug: BI 44370 tablet; Other: high fat breakfast

INTERVENTIONS:
Drug: BI 44370 powder for oral solution
  Arms: Treatment A; Treatment B; Treatment C; Treatment D
Drug: BI 44370 tablet
  Arms: Treatment E; Treatment F
Other: high fat breakfast
  Arms: Treatment B; Treatment D; Treatment F

SUMMARY:
The objective of this trial was to evaluate the relative oral bioavailability and pharmacokinetics of BI 44370 TA drinking solution (100 mg and 200 mg) and BI 44370 TA tablets (100 mg as two 50 mg tablets) with and without a high fat meal and to assess the safety and tolerability of the substances.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects according to the following criteria based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥21 and ≤55 years
* BMI ≥18.5 and ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR, and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family, history of Long QT Syndrome)

For Male Subjects:

* Not willing to use adequate contraception (condoms use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole study period from the time of the first intake of study drug until three months after the last intake

For Female Subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception e.g. sterilisation, intrauterine pessary (IUP), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period during the whole study period from the time of the first intake of study drug until one month after the last intake
* Lactation period

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | up to 24 hours after drug administration
AUC0-2 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 2 h after drug administration) | up to 2 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours after drug administration
tmax (time from dosing to maximum measured concentration) | up to 24 hours after drug administration

SECONDARY OUTCOMES:
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 24 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 24 hours after drug administration
AUCt1-t2 (Area under the concentration-time curve of the analyte in plasma over the time interval t1 to t2) | up to 24 hours after drug administration
λz (terminal rate constant in plasma) | up to 24 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 24 hours after drug administration
MRTp.o. (mean residence time of the analyte in the body after p.o. administration) | up to 24 hours after drug administration
CL/F (total/apparent clearance of the analyte in plasma after extravascular administration) | up to 24 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 24 hours after drug administration
Number of patients with clinically relevant findings in vital signs (blood pressure and pulse rate) | up to 11 days
Number of patients with clinically relevant findings in 12-lead ECG (electrocardiogram) | up to 11 days
Number of patients with clinically relevant laboratory findings | up to 11 days
Number of patients with adverse events | up to 34 days
Assessment of tolerability by investigator on a 4-point scale | within 10 days after administration of study drug